CLINICAL TRIAL: NCT06042816
Title: Evaluation of the Analgesic Efficacy of Free Opioid Anesthesia for Patients Undergoing Colectomies and Rectal Resections: A Prospective, Randomized Controlled Clinical Trial
Brief Title: Analgesic Efficacy of Free-opioid Anesthesia for Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vietnam Military Medical University (Other)
Responsible Party: Principal Investigator, Nguyen Trung Kien, Assoc. Prof, Nguyen Trung Kien, PhD, MD. Director of Center of Emergency, Critical Care Medicine and Clinical Toxicology, Military Hospital 103, Vietnam Military Medical University, Vietnam, Vietnam Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 01/CN-HDĐ
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Cancer
Keywords: Free-opioid anesthesia; Opioid anesthesia; colorectal surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients were randomized into 2 groups: Group OA - Opioid anesthesia (n = 49): Intraoperative pain control by fentanyl; FOA group - Free-opioid anesthesia (n = 49): Intraoperative pain control by continuous infusion of lidocaine, bolus doses of ketamine combined with epidural levobupivacaine.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The drugs were administered in 10 mL and 50 mL syringes labeled as ''loading'' or ''infusion'' respectively. All the drugs delivered in loading dose (intravenous lidocaine and ketamine, epidural levobupivacaine in FOA group; fentanyl and normal saline in OA group) were diluted in normal saline to 10 ml volume labeled indistinguishably as ''loading-1'' and ''loading-2'', "loading-3"…. Because the number of loading drugs in the FOA group was greater than in OA group, investigators added some 10 ml normal saline syringes in the OA group to make the number of "loading" syringes in the two groups equal, thereby ensuring complete blinding. The infusion drugs (lidocaine, ketamine and levobupivacaine in FOA group or normal saline in OA group) were prepared in 50 mL syringes and labeled as ''infusion-1'' and''infusion-2'' respectively. The patients and the anesthetists taking part in the procedures were not informed of the study protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free-opioid anesthesia (Experimental): 49 patients were injected bolus doses of lidocaine 1 mg/kg and ketamine 0.5 mg/kg before induction. Then intravenous propofol 1% 2-2.5 mg/kg, rocuronium 0.6 mg/kg were utilized for induction. For anesthesia maintenance, patients received intraoperative multimodal analgesia, in which an epidural bolus of 3 - 5 ml of levobupivacaine 0.1% was followed by a continuous infusion of 3 - 5 ml/h epidurally; in addition, intravenous infusion of lidocaine 1 mg/kg/hour and ketamine 0.25 mg/kg/h were maintained until the end of surgery. Patients were given a bolus of 3-5 ml levobupivacaine 0.1% epidurally and ketamine 0.25 mg/kg intravenously if SPI > 50, 40 < SE < 60, TOF = 0 and hemodynamics was stable. Postoperative pain management was implemented with patient-controlled epidural levobupivacaine 0.1% for 72 hours, and pain rescue with fentanyl 0.5 μg/kg.
  Interventions: Procedure: Free-opioid anesthesia
- Opioid anesthesia (Active Comparator): 49 patients received a bolus dose of fentanyl 2 µg/kg before induction of anesthesia. For anesthesia maintenance, in group OA, a bolus dose of fentanyl 3 µg/kg was given 5 minutes before skin incision, and then a continuous infusion of fentanyl 2 µg/kg/h was maintained for intraoperative pain management; fentanyl 0.5 μg/kg was bolused when SPI (Surgical Pleth Index) > 50, 40 < State Entropy (SE) < 60, Train of four (TOF) = 0 and the patient was hemodynamically stable. Propofol and fentanyl were discontinued at the start of skin closure. Postoperative pain management was implemented with patient-controlled epidural levobupivacaine 0.1% for 72 hours, and pain rescue with fentanyl 0.5 μg/kg.
  Interventions: Procedure: opioid anesthesia

INTERVENTIONS:
Procedure: Free-opioid anesthesia — Free opioid anesthesia (FOA) has been used in many countries around the world, making use of multimodal analgesia therapy which includes hypnotics, N-methyl-D-aspartate (NMDA) antagonists, local anesthetics and anti-inflammatory agents and sympathetic block in surgery. This method was demonstrated to contribute to enhanced recovery after surgery (ERAS). The use of long-acting local anesthetics also enhances postoperative pain relief. As a result, the concept of balanced anesthesia now has a change in three basic components: hypnotics, muscle relaxants and sympathomimetic inhibitors
  Arms: Free-opioid anesthesia
Procedure: opioid anesthesia — Opioids have been used as one of three basic components of balanced anesthesia, including anesthetic drugs, pain relievers, and neuromuscular blockade agents (opioid anesthesia). Opioids not only facilitate deep anesthesia but also create the most favorable conditions for surgeries. Fentanyl is a potent opioid used to control pain, reduce the dose of sympathomimetic inhibitors and maintain hemodynamic stability. However, several common side effects of fentanyl are well known: nausea and vomiting, constipation, urinary retention, headache, pruritus, rash, histamine release, biliary spasm and respiratory depression, the most severe adverse effect
  Arms: Opioid anesthesia

SUMMARY:
Objectives: To compare free-opioid anesthesia (the combination of epidural anesthesia, intravenous lidocaine, ketamine, propofol, and sevoflurane) and opioid anesthesia (fentanyl, propofol and sevoflurane) regarding intraoperative analgesic efficacy in colectomies and rectal resections at Viet Tiep Friendship Hospital.

Methods: A prospective, randomized controlled clinical trial was performed on 98 patients who were anesthetized for colorectal surgery from December 2019 to November 2021. Patients were randomized into 2 groups: Group OA - Opioid anesthesia (n = 49): Intraoperative pain control by fentanyl; FOA group - Free-opioid anesthesia (n = 49): Intraoperative pain control by continuous infusion of lidocaine, bolus doses of ketamine combined with epidural levobupivacaine.

DETAILED DESCRIPTION:
After being placed an epidural catheter and given a bolus dose of dexamethasone 0.1 mg/kg, patients was endotracheal anesthetized with propofol 1% 2-2.5 mg/kg, rocuronium 0.6 mg/kg. Intubation was implemented when TOF (Train Of Four)=0 and RE (Response Entropy), SE (State Entropy) ≤ 60. Patients in OA group received a bolus dose of fentanyl 2 µg/kg before induction of anesthesia while those in FOA group received bolus doses of lidocaine 1 mg/kg and ketamine 0.5 mg/kg. In FOA group, lidocaine 10% was sprayed on the patients glottis to facilitate intubation.

For anesthesia maintenance, in group OA, a bolus dose of fentanyl 3 µg/kg was given 5 minutes before skin incision, and then a continuous infusion of fentanyl 2 µg/kg/h was maintained for intraoperative pain management; fentanyl 0.5 μg/kg was bolused when SPI (Surgical Pleth Index) > 50, 40 < SE < 60, TOF = 0 and the patient was hemodynamically stable. Propofol and fentanyl were discontinued at the start of skin closure. In FOA group, patients received intraoperative multimodal analgesia, in which an epidural bolus of 3 - 5 ml of levobupivacaine 0.1% was followed by a continuous infusion of 3 - 5 ml/h epidurally; in addition, intravenous infusion of lidocaine 1 mg/kg/hour and ketamine 0.25 mg/kg/h were maintained until the end of surgery. Patients were given a bolus of 3-5 ml levobupivacaine 0.1% epidurally and ketamine 0.25 mg/kg intravenously if SPI > 50, 40 < SE < 60, TOF = 0 and hemodynamics was stable.

For all patients, anesthesia was maintained by volatile anesthetics (Sevoflurane or Desflurane) to ensure 40 < SE < 60, and rocuronium 0.2 mg/kg was repeated when TOF = 2 (the last injection of neuromuscular blockade was not given when the estimated duration from the point of injection to the point of abdominal closure is shorter than 20 minutes). Mechanical ventilation was provided with a tidal volume 6-8 ml/kg in the volume-controlled mode and respiratory rate at 10-12 breath/minute, FiO2 (Fraction of inspired oxygen)=50%. Peak airway pressure was maintained within the range of 12-16 cmH2O and EtCO2 (End-tidal Carbon dioxide) was kept from 35 to 40 mmHg with a fresh gas flow of 1.2 - 2 liters/minute. At the end of surgery, reversal of neuromuscular blockade was performed with neostigmine combined with atropine, and extubation was carried out when patients met the criteria. Postoperative pain management was implemented with patient-controlled epidural levobupivacaine 0.1% for 72 hours, and pain rescue with fentanyl 0.5 μg/kg.

ELIGIBILITY:
Inclusion Criteria:

* Patients agreed to participate in the study.
* Patients aged ≥ 18 years old,
* Those who underwent elective colectomies or rectal resections,
* Those who were ASA (American Society of Anesthesiologists) classified as I - III,
* Those who were indicated for general endotracheal anesthesia from December 2019 to November 2021 at Viet Tiep Friendship Hospital

Exclusion Criteria:

* Patients refused to participate in the study,
* Patients had BMI (Body Mass Index) ≥ 35;
* Pregnant or lactating or menstruating women;
* Those who had liver failure, renal failure, heart failure, history of chronic pain, alcohol or drug abuse, mental illnesses, allergies or contraindications to any studied medications.
* Those who were unable to assess pain or use of patient-controlled analgesia devices (PCA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
analgesic efficacy of free-opioid anesthesia | before induction of anesthesia
  intraoperative alteration of Surgical Pleth Index (SPI). The Surgical Pleth Index (SPI) is an objective tool that can reflect nociception-antinociception balance and guide the use of intraoperative analgesics. The values of the SPI range from 0 to 100. During general anaesthesia, maintaining a value between 20 and 50 is generally recommended. When the SPI value is greater than 50 and exceeds 3-5 min, it routinely indicates that the noxious stimulation is too strong and that additional analgesic drugs are needed.
analgesic efficacy of free-opioid anesthesia | After intubation
  intraoperative alteration of Surgical Pleth Index (SPI)
analgesic efficacy of free-opioid anesthesia | After skin incision
  intraoperative alteration of Surgical Pleth Index (SPI)
analgesic efficacy of free-opioid anesthesia | when the restoration of eyelids reflex emerged
  intraoperative alteration of Surgical Pleth Index (SPI)
analgesic efficacy of free-opioid anesthesia | Intraoperatively (From the induction of anesthesia to the emergence)
  The number of times of intraoperative analgesics adjustment
analgesic efficacy of free-opioid anesthesia | postoperatively (upto 3 days after surgery)
  the proportion of patients requiring postoperative pain rescue

SECONDARY OUTCOMES:
Effects of free-opioid anesthesia on intraoperative mean arterial blood pressure | T0 (right after entering the operating theatre)
  Non-invasive blood pressure was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The mean arterial blood pressure at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative mean arterial blood pressure | T1 (before induction of anesthesia)
  Non-invasive blood pressure was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The mean arterial blood pressure at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative mean arterial blood pressure | T2 (patients lost eyelid reflex and response to verbal command)
  Non-invasive blood pressure was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The mean arterial blood pressure at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative mean arterial blood pressure | T3 (before intubation)
  Non-invasive blood pressure was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The mean arterial blood pressure at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative mean arterial blood pressure | T4 (after intubation)
  Non-invasive blood pressure was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The mean arterial blood pressure at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative mean arterial blood pressure | T5 (before skin incision)
  Non-invasive blood pressure was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The mean arterial blood pressure at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative mean arterial blood pressure | T6 (after skin incision)
  Non-invasive blood pressure was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The mean arterial blood pressure at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative mean arterial blood pressure | T7 (colon release)
  Non-invasive blood pressure was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The mean arterial blood pressure at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative mean arterial blood pressure | T8 (dissection of colorectal mesentery)
  Non-invasive blood pressure was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The mean arterial blood pressure at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative mean arterial blood pressure | T9 (colon resection)
  Non-invasive blood pressure was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The mean arterial blood pressure at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative mean arterial blood pressure | T10 (restore gastrointestinal flow)
  Non-invasive blood pressure was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The mean arterial blood pressure at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative mean arterial blood pressure | T11 (drainage placement)
  Non-invasive blood pressure was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The mean arterial blood pressure at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative mean arterial blood pressure | T12 (before skin closure)
  Non-invasive blood pressure was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The mean arterial blood pressure at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative mean arterial blood pressure | T13 (immediately after skin closure)
  Non-invasive blood pressure was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The mean arterial blood pressure at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative mean arterial blood pressure | T14 (eyelids reflex restored and patients eyes could open on command)
  Non-invasive blood pressure was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The mean arterial blood pressure at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative mean arterial blood pressure | T15 (before extubation)
  Non-invasive blood pressure was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The mean arterial blood pressure at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative mean arterial blood pressure | T16 (15 minutes after extubation)
  Non-invasive blood pressure was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The mean arterial blood pressure at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative heart rate | T0 (right after entering the operating theatre)
  Heart rate was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The heart rate at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative heart rate | T1 (before induction of anesthesia)
  Heart rate was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The heart rate at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative heart rate | T2 (patients lost eyelid reflex and response to verbal command)
  Heart rate was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The heart rate at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative heart rate | T3 (before intubation)
  Heart rate was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The heart rate at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative heart rate | T4 (after intubation)
  Heart rate was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The heart rate at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative heart rate | T5 (before skin incision)
  Heart rate was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The heart rate at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative heart rate | T6 (after skin incision)
  Heart rate was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The heart rate at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative heart rate | T7 (colon release)
  Heart rate was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The heart rate at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative heart rate | T8 (dissection of colorectal mesentery)
  Heart rate was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The heart rate at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative heart rate | T9 (colon resection)
  Heart rate was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The heart rate at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative heart rate | T10 (restore gastrointestinal flow)
  Heart rate was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The heart rate at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative heart rate | T11 (drainage placement)
  Heart rate was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The heart rate at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative heart rate | T12 (before skin closure)
  Heart rate was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The heart rate at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative heart rate | T13 (immediately after skin closure)
  Heart rate was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The heart rate at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative heart rate | T14 (eyelids reflex restored and patients eyes could open on command)
  Heart rate was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The heart rate at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative heart rate | T15 (before extubation)
  Heart rate was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The heart rate at each time point was compared between the two groups.
Effects of free-opioid anesthesia on intraoperative heart rate | T16 (15 minutes after extubation)
  Heart rate was assessed every 5 minutes intraoperatively and recorded at some investigated time points. The heart rate at each time point was compared between the two groups.
changes in the concentration of IL (Interleukin)-6 | Before surgery
  Blood samples were collected in a heparin tube immediately before surgery (T0) and 1 hour after extubation. They were centrifuged, and then plasma was separated and stored at -70°C until being analyzed. IL-6 levels were analyzed using enzyme-linked immunosorbent assay (ELISA). Changes in IL-6 were recorded and compared between the two groups
changes in the concentration of IL (Interleukin)-6 | 1 hour after surgery
  Blood samples were collected in a heparin tube immediately before surgery (T0) and 1 hour after extubation. They were centrifuged, and then plasma was separated and stored at -70°C until being analyzed. IL-6 levels were analyzed using enzyme-linked immunosorbent assay (ELISA). Changes in IL-6 were recorded and compared between the two groups
changes in the concentration of IL-10 | Before surgery
  Blood samples were collected in a heparin tube immediately before surgery (T0) and 1 hour after extubation. They were centrifuged, and then plasma was separated and stored at -70°C until being analyzed. IL-10 levels were analyzed using enzyme-linked immunosorbent assay (ELISA). Changes in IL-10 were recorded and compared between the two groups
changes in the concentration of IL-10 | 1 hour after surgery
  Blood samples were collected in a heparin tube immediately before surgery (T0) and 1 hour after extubation. They were centrifuged, and then plasma was separated and stored at -70°C until being analyzed. IL-10 levels were analyzed using enzyme-linked immunosorbent assay (ELISA). Changes in IL-10 were recorded and compared between the two groups
Adverse effects of free-opioid anesthesia | up to 3 days postoperatively
  the rate of patients suffering nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Kien T Nguyen, Ph.D, Study Director — Center of Emergency, Critical Care Medicine and Clinical Toxicology, Military Hospital 103, Vietnam
Locations (1):
- Viet-Tiep Friendship Hospital, Haiphong, Le Chan, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during this study are available from the corresponding author on reasonable request. Researchers could contact the corresponding author via email to ask for IPD.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available when the publication is completed
Access Criteria: The data is available only for research purposes and personal information of the participants need to be kept confidential

REFERENCES:
- [Result] Vaswani JP, Debata D, Vyas V, Pattil S. Comparative Study of the Effect of Dexmedetomidine Vs. Fentanyl on Haemodynamic Response in Patients Undergoing Elective Laparoscopic Surgery. J Clin Diagn Res. 2017 Sep;11(9):UC04-UC08. doi: 10.7860/JCDR/2017/27020.10578. Epub 2017 Sep 1. PMID 29207810
- [Result] Choi H, Song JY, Oh EJ, Chae MS, Yu S, Moon YE. The Effect of Opioid-Free Anesthesia on the Quality of Recovery After Gynecological Laparoscopy: A Prospective Randomized Controlled Trial. J Pain Res. 2022 Aug 3;15:2197-2209. doi: 10.2147/JPR.S373412. eCollection 2022. PMID 35945992
- [Result] Bakan M, Umutoglu T, Topuz U, Uysal H, Bayram M, Kadioglu H, Salihoglu Z. Opioid-free total intravenous anesthesia with propofol, dexmedetomidine and lidocaine infusions for laparoscopic cholecystectomy: a prospective, randomized, double-blinded study. Braz J Anesthesiol. 2015 May-Jun;65(3):191-9. doi: 10.1016/j.bjane.2014.05.001. Epub 2014 Jun 3. PMID 25925031
- [Result] Hakim KYK, Wahba WZB. Opioid-Free Total Intravenous Anesthesia Improves Postoperative Quality of Recovery after Ambulatory Gynecologic Laparoscopy. Anesth Essays Res. 2019 Apr-Jun;13(2):199-203. doi: 10.4103/aer.AER_74_19. PMID 31198230
- [Result] Chin KJ, Lewis S. Opioid-free Analgesia for Posterior Spinal Fusion Surgery Using Erector Spinae Plane (ESP) Blocks in a Multimodal Anesthetic Regimen. Spine (Phila Pa 1976). 2019 Mar 15;44(6):E379-E383. doi: 10.1097/BRS.0000000000002855. PMID 30180150